CLINICAL TRIAL: NCT01709500
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of REGN727/SAR236553 in Patients With Heterozygous Familial Hypercholesterolemia Not Adequately Controlled With Their Lipid-Modifying Therapy
Brief Title: Study of Alirocumab (REGN727/SAR236553) in Patients With heFH (Heterozygous Familial Hypercholesterolemia) Who Are Not Adequately Controlled With Their LMT (Lipid-Modifying Therapy)
Acronym: ODYSSEY FH II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R727-CL-1112
Record Dates: First submitted 2012-10-08; First posted 2012-10-18 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-09

CONDITIONS: Heterozygous Familial Hypercholesterolemia
MeSH Terms: interventions — Atorvastatin; Simvastatin; Rosuvastatin Calcium; alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alirocumab 75 mg/up to 150 mg (Experimental): Alirocumab 75 mg every two weeks (Q2W) added to stable dose of statin with or without LMT for 78 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL at Week 8.
  Interventions: Drug: LMT (atorvastatin, simvastatin, or rosuvastatin); Drug: alirocumab
- Placebo (Placebo Comparator): Placebo matched to alirocumab SC injection for 78-week treatment duration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LMT (atorvastatin, simvastatin, or rosuvastatin)
  Arms: Alirocumab 75 mg/up to 150 mg
Drug: alirocumab — Alirocumab administered as a subcutaneous (SC) injection of 1 mL into the abdomen, thigh, or outer area of the upper arm.
  Other Names: REGN727; SAR236553
  Arms: Alirocumab 75 mg/up to 150 mg
Drug: Placebo — Placebo matched to alirocumab administered as a SC injection of 1 mL into the abdomen, thigh, or outer area of the upper arm.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, multi-national study alirocumab (REGN727/SAR236553) in patients with Heterozygous Familial Hypercholesterolemia (heFH) who are not adequately controlled with their Lipid-Modifying Therapy (LMT).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with heFH* who are not adequately controlled** with a maximally-tolerated daily dose*** of statin with or without other LMT, at a stable dose prior to the screening visit (week -2).

   *Diagnosis of heFH must be made either by genotyping or by clinical criteria. For those patients not genotyped, the clinical diagnosis may be based on either the Simon Broome criteria for definite FH (Appendix 1) or the WHO/Dutch Lipid Network criteria with a score of >8 points (Appendix 2).

   ** "Not adequately controlled" is defined as LDL-C ≥70 mg/dL (1.81 mmol/L) at the screening visit (week -2) in patients with a history of documented CVD (Appendix 3), or LDL-C ≥100 mg/dL (2.59 mmol/L) at the screening visit (week -2) in patients without a history of documented CVD.

   *** "Maximally-tolerated dose" is defined as (any of the following are acceptable):
   * Rosuvastatin 20 mg or 40 mg daily
   * Atorvastatin 40 mg or 80 mg daily
   * Simvastatin 80 mg daily (if already on this dose for >1 year - see exclusion criterion #7)

   Note: Patients who are not able to be on any of the above statin doses should be treated with the dose of daily atorvastatin, rosuvastatin, or simvastatin which is considered appropriate for the patient, according to the investigator's judgment. Some examples of acceptable reasons for a patient taking a lower statin dose include, but are not limited to: adverse effects on higher doses, advanced age, low body mass index, regional practices, local prescribing information, concomitant medications, co-morbid conditions such as impaired glucose tolerance/impaired fasting glucose. The reason(s) will be documented in the case report form (CRF).
2. Provide signed informed consent

Exclusion Criteria:

1. Patient without diagnosis of heFH made either by genotyping or by clinical criteria
2. LDL-C <70 mg/dL (<1.81 mmol/L) at the screening visit (week-2) in patients with history of documented cardiovascular disease
3. LDL-C <100 mg/dL (<2.59 mmol/L) at the screening visit (week -2) in patients without history of documented cardiovascular disease
4. Not on a stable dose of LMT (including statin) for at least 4 weeks and/or fenofibrate for at least 6 weeks, as applicable, prior to the screening visit (week -2) and from screening to randomization
5. Currently taking another statin than simvastatin, atorvastatin, or rosuvastatin
6. Simvastatin, atorvastatin, or rosuvastatin is not taken daily or not taken at a registered dose
7. Daily doses above atorvastatin 80 mg, rosuvastatin 40 mg, or simvastatin 40 mg (except for patients on simvastatin 80 mg for more than 1 year, who are eligible)
8. Use of fibrates, other than fenofibrate within 6 weeks of the screening visit (week-2) or between screening and randomization visits
9. Use of nutraceutical products or over-the-counter therapies that may affect lipids which have not been at a stable dose/amount for at least 4 weeks prior to the screening visit (week -2) or between screening and randomization visits
10. Use of red yeast rice products within 4 weeks of the screening visit (week-2), or between screening and randomization visits
11. Patient who has received plasmapheresis treatment within 2 months prior to the screening visit (week -2), or has plans to receive it during the study
12. Recent (within 3 months prior to the screening visit [week -2] or between screening and randomization visits) MI, unstable angina leading to hospitalization, percutaneous coronary intervention (PCI), coronary artery bypass graft surgery (CABG), uncontrolled cardiac arrhythmia, stroke, transient ischemic attack (TIA), carotid revascularization, endovascular procedure or surgical intervention for peripheral vascular disease

(The inclusion/exclusion criteria provided above is not intended to contain all considerations relevant to a participant's potential participation in this clinical trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2012-12; Primary Completion 2014-05 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (24):
- Czechia (4):
  - Hradec Králové
  - Prague
  - Trutnov
  - Vyškov
- Netherlands (13):
  - Alkmaar
  - Amsterdam
  - Apeldoorn
  - Enschede
  - Goes
  - Groningen
  - Hoogeveen
  - Hoorn
  - Rotterdam
  - Sittard- Geleen
  - Utrecht (2 Locations)
  - Venlo
  - Waalwijk
- Oslo, Norway
- United Kingdom (6):
  - Cardiff
  - London
  - Manchester
  - Middlesex
  - Newcastle upon Tyne
  - West Bromwich

REFERENCES:
- [Derived] Mahmood T, Minnier J, Ito MK, Li QH, Koren A, Kam IW, Fazio S, Shapiro MD. Discordant responses of plasma low-density lipoprotein cholesterol and lipoprotein(a) to alirocumab: A pooled analysis from 10 ODYSSEY Phase 3 studies. Eur J Prev Cardiol. 2021 Jul 23;28(8):816-822. doi: 10.1177/2047487320915803. Epub 2020 Apr 10. PMID 34298554
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102
- [Derived] Defesche JC, Stefanutti C, Langslet G, Hopkins PN, Seiz W, Baccara-Dinet MT, Hamon SC, Banerjee P, Kastelein JJP. Efficacy of alirocumab in 1191 patients with a wide spectrum of mutations in genes causative for familial hypercholesterolemia. J Clin Lipidol. 2017 Nov-Dec;11(6):1338-1346.e7. doi: 10.1016/j.jacl.2017.08.016. Epub 2017 Sep 4. PMID 28964736
- [Derived] Kastelein JJ, Hovingh GK, Langslet G, Baccara-Dinet MT, Gipe DA, Chaudhari U, Zhao J, Minini P, Farnier M. Efficacy and safety of the proprotein convertase subtilisin/kexin type 9 monoclonal antibody alirocumab vs placebo in patients with heterozygous familial hypercholesterolemia. J Clin Lipidol. 2017 Jan-Feb;11(1):195-203.e4. doi: 10.1016/j.jacl.2016.12.004. Epub 2016 Dec 28. PMID 28391886
- [Derived] Ray KK, Ginsberg HN, Davidson MH, Pordy R, Bessac L, Minini P, Eckel RH, Cannon CP. Reductions in Atherogenic Lipids and Major Cardiovascular Events: A Pooled Analysis of 10 ODYSSEY Trials Comparing Alirocumab With Control. Circulation. 2016 Dec 13;134(24):1931-1943. doi: 10.1161/CIRCULATIONAHA.116.024604. Epub 2016 Oct 24. PMID 27777279
- [Derived] Kastelein JJ, Ginsberg HN, Langslet G, Hovingh GK, Ceska R, Dufour R, Blom D, Civeira F, Krempf M, Lorenzato C, Zhao J, Pordy R, Baccara-Dinet MT, Gipe DA, Geiger MJ, Farnier M. ODYSSEY FH I and FH II: 78 week results with alirocumab treatment in 735 patients with heterozygous familial hypercholesterolaemia. Eur Heart J. 2015 Nov 14;36(43):2996-3003. doi: 10.1093/eurheartj/ehv370. Epub 2015 Sep 1. PMID 26330422
- [Derived] Kastelein JJ, Robinson JG, Farnier M, Krempf M, Langslet G, Lorenzato C, Gipe DA, Baccara-Dinet MT. Efficacy and safety of alirocumab in patients with heterozygous familial hypercholesterolemia not adequately controlled with current lipid-lowering therapy: design and rationale of the ODYSSEY FH studies. Cardiovasc Drugs Ther. 2014 Jun;28(3):281-9. doi: 10.1007/s10557-014-6523-z. PMID 24842558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 26 sites in 4 countries. Overall, 322 participants were screened between 28 Nov 2012 and 26 Apr 2013, 73 of whom were screen failures.
Pre-assignment Details: Randomization was stratified according to prior history of myocardial infarction or ischemic stroke, and intensity of statin treatment. Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 2:1 (alirocumab: placebo) ratio after confirmation of selection criteria.
Groups:
- Alirocumab 75 mg/up to 150 mg: Alirocumab 75 mg SC injection every two weeks (Q2W) added to stable dose of statin with or without LMT for 78 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL at Week 8.
Period: Overall Study
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Started | 167 | 82
Treated | 167 | 81
Completed | 0 | 0
Not Completed | 167 | 82
Not completed — Randomized but not treated | 0 | 1
Not completed — Adverse Event | 5 | 1
Not completed — Poor compliance to protocol | 2 | 1
Not completed — Other | 3 | 1
Not completed — Related to IMP administration | 1 | 0
Not completed — Treatment ongoing | 156 | 78

BASELINE CHARACTERISTICS:
Groups:
- Alirocumab 75 mg/up to 150 mg: Alirocumab 75 mg SC injection Q2W added to stable dose of statin with or without LMT for 78 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL at Week 8.
- Placebo: Placebo matched to alirocumab SC injection for 78--week treatment duration.
- Total: Total of all reporting groups
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo | Total
Number analyzed (Participants) | 167 | 82 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (12.93) | 53.2 (12.55) | 53.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 37 | 118
  Male | 86 | 45 | 131
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] — Calculated LDL-C values were obtained using Friedewald formula.
  mmol/L | 3.485 (1.065) | 3.471 (1.071) | 3.480 (1.065)
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C values were obtained using Friedewald formula.
  mg/dL | 134.6 (41.1) | 134.0 (41.4) | 134.4 (41.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - Intent--to--Treat (ITT) Analysis
Description: Calculated LDL-C values were obtained using the Friedewald formula. Adjusted Least- squares (LS) means and standard errors at Week 24 were obtained from a mixed -effect model with repeated measures (MMRM) to account for missing data. All available post -baseline data from Week 4 to Week 52 regardless of status on- or off-treatment were used in the model.
Time Frame: From Baseline to Week 52
Population: ITT population: all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -48.7 (1.9) | 2.8 (2.8)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Alirocumab group was compared to the placebo group using an appropriate contrast statement; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -51.4, 95% CI 2-sided [-58.1 to -44.8]

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - On-Treatment Analysis
Description: Calculated LDL-C values were obtained using the Friedewald formula. Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection) (on-treatment analysis).
Time Frame: From Baseline to Week 52
Population: Modified ITT (mITT) population: all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -49.4 (1.9) | 2.7 (2.7)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 5% level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -52.2, 95% CI 2-sided [-58.7 to -45.6]

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment (ITT analysis).
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -43.8 (1.8) | 4.6 (2.6)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -48.4, 95% CI 2-sided [-54.7 to -42.2]

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On- Treatment Analysis
Description: Calculated LDL-C values were obtained using the Friedewald formula. Adjusted LS means and standard errors at Week 12 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection) (on-treatment analysis).
Time Frame: From Baseline to Week 52
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -44.2 (1.8) | 4.6 (2.6)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -48.8, 95% CI 2-sided [-55 to -42.5]

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 163 | 81
percent change | -42.8 (1.4) | -3.5 (2)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -39.3, 95% CI 2-sided [-44.1 to -34.5]

6. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 52
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 162 | 80
percent change | -43.2 (1.4) | -3.5 (2)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -39.8, 95% CI 2-sided [-44.5 to -35.1]

7. Secondary Outcome: Percent Change From Baseline in Non-High -Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 52
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -42.6 (1.8) | 3.1 (2.5)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -45.7, 95% CI 2-sided [-51.8 to -39.7]

8. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 - On-Treatment Analysis
Description: as for outcome 6
Time Frame: From Baseline to Week 52
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -43.2 (1.7) | 3.1 (2.5)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -46.4, 95% CI 2-sided [-52.3 to -40.4]

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 52
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline total-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -30.6 (1.4) | 2.1 (1.9)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean difference = -32.8, 95% CI 2-sided [-37.4 to -28.1]

10. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: Apo B ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 163 | 81
percent change | -35.4 (1.4) | -0.9 (2)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -34.5, 95% CI 2-sided [-39.2 to -29.8]

11. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 52
Population: Non-HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -37.9 (1.7) | 4.1 (2.4)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -42, 95% CI 2-sided [-47.8 to -36.2]

12. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post baseline data from Week 4 to Week 52 regardless of status on- or off treatment.
Time Frame: From Baseline to Week 52
Population: Total--C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -26.6 (1.3) | 3.4 (1.9)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Threshold for significance ≤ 0.05; LS Mean Difference = -29.9, 95% CI 2-sided [-34.5 to -25.4]

13. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 52 - ITT Analysis
Description: Calculated LDL-C values were obtained using the Friedewald formula. Adjusted LS means and standard errors at Week 52 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on- or off treatment (ITT analysis).
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -50.3 (2.3) | 8.4 (3.3)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -58.8, 95% CI 2-sided [-66.8 to -50.8]

14. Secondary Outcome: Percentage of Very High CV Risk Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) or High CV Risk Participants Reaching Calculated LDL-C <100 mg/dL (2.59 mmol/L) at Week 24 - ITT Analysis
Description: Adjusted percentages at Week 24 were obtained from a multiple imputation approach model for handling of missing data. All available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment were included in the imputation model (ITT analysis).
Time Frame: Up to Week 52
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percentage of participants | 81.4 | 11.3
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant). Statistical analysis used a multiple imputation approach followed by a Logistic regression model; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Odds Ratio (OR) = 52.2, 95% CI 2-sided [20.9 to 130]

15. Secondary Outcome: Percentage of Very High CV Risk Participants Reaching Calculated LDL--C <70 mg/dL (1.81 mmol/L) or High CV Risk Participants Reaching Calculated LDL--C <100 mg/dL (2.59 mmol/L) at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 were obtained from a multiple imputation approach model including available post-baseline on-treatment data from Week 4 to Week 52 i.e. up to 21 days after last injection (on-treatment analysis).
Time Frame: Up to week 52
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percentage of participants | 82.1 | 11.6
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Odds Ratio (OR) = 53.3, 95% CI 2-sided [21.4 to 132.6]

16. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - ITT Analysis
Description: as for outcome 14
Time Frame: Up to Week 52
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percentage of participants | 68.2 | 1.2
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Odds Ratio (OR) = 239.7, 95% CI 2-sided [31.6 to 1820.3]

17. Secondary Outcome: Percentage of Participants Reaching Calculated LDL--C <70 mg/dL (1.81 mmol/L) at Week 52 - On-Treatment Analysis
Description: Adjusted percentages at Week 52 were obtained from a multiple imputation approach model including available post-baseline on-treatment data from Week 4 to Week 52 i.e. up to 21 days after last injection (on-treatment analysis).
Time Frame: Up to Week 52
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percentage of participants | 68.8 | 1.3
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Odds Ratio (OR) = 240.6, 95% CI 2-sided [31.4 to 1841.7]

18. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from a multiple imputation approach model including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: Participants analyzed: participants of the ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -30.3 (1.8) | -10 (2.5)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant). Statistical analysis used a multiple imputation approach followed by a robust regression model; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Adjusted Mean Difference = -20.3, 95% CI 2-sided [-26.4 to -14.2]

19. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | 6.0 (1.2) | -0.8 (1.6)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 6.8, 95% CI 2-sided [2.8 to 10.7]

20. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: as for outcome 18
Time Frame: From Baseline to Week 52
Population: Participants analyzed: participants of the ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -10.4 (2) | 0.5 (2.8)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure. Statistical analysis used a multiple imputation approach followed by a robust regression model; Test type: Superiority or Other; p = 0.0012, Regression, Robust — Threshold for significance ≤ 0.05; Adjusted Mean Difference = -10.9, 95% CI 2-sided [-17.5 to -4.3]

21. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 24 - ITT Analysis
Description: as for outcome 19
Time Frame: From Baseline to Week 52
Population: Participants analyzed: participants of the ITT population with one baseline and at least one post-baseline Apo A-1 value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 163 | 81
percent change | 2.8 (0.9) | -1.6 (1.3)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p = 0.0062, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 4.4, 95% CI 2-sided [1.3 to 7.5]

22. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 from a multiple imputation approach model including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: Lipoprotein (a) ITT population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -24.7 (1.7) | -5.6 (2.5)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Adjusted Mean Difference = -19.1, 95% CI 2-sided [-25 to -13.1]

23. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 52 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 52
Population: HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | 6.0 (1.0) | -0.8 (1.6)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p = 0.0147, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 4.3, 95% CI 2-sided [0.9 to 7.8]

24. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 12 - ITT Analysis
Description: as for outcome 22
Time Frame: From Baseline to Week 52
Population: Fasting triglycerides ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 166 | 81
percent change | -8.1 (2.2) | 0.6 (3.1)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.024, Regression, Robust — Threshold for significance ≤ 0.05; Adjusted Mean Difference = -8.6, 95% CI 2-sided [-16.1 to -1.1]

25. Secondary Outcome: Percent Change From Baseline in Apo A-1 at Week 12 - ITT Analysis
Description: as for outcome 23
Time Frame: From Baseline to Week 52
Population: Apo A-1 ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Number analyzed (Participants) | 163 | 81
percent change | 0.4 (0.9) | -1.9 (1.3)
Statistical Analysis 1: Comparison: Alirocumab 75 mg/up to 150 mg vs Placebo; Testing according to the hierarchical testing procedure (previous endpoints were statistically significant); Test type: Superiority or Other; p = 0.1475, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 2.3, 95% CI 2-sided [-0.8 to 5.5]

ADVERSE EVENTS:
Time Frame: From Baseline up to Week 78
Description: Treatment emergent adverse events that developed during treatment emergent adverse events period (the time from the first dose of study drug to the last dose of study drug + 70 days (10 weeks) are reported.
Groups:
- Alirocumab 75 mg/up to 150 mg: Alirocumab 75 mg SC injection every two weeks (Q2W) added to stable dose of statin with or without LMT for 76 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when LDL-C levels ≥70 mg/dL at Week 8.
Arm/Group | Alirocumab 75 mg/up to 150 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 10/167 | 7/81
Other Adverse Events (participants affected / at risk) | 65/167 | 35/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alirocumab 75 mg/up to 150 mg (N=167) | Placebo (N=81)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Device dislocation (General disorders) | 1 | 0
Non-Cardiac chest pain (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Hepatitis a (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alirocumab 75 mg/up to 150 mg (N=167) | Placebo (N=81)
Diarrhoea (Gastrointestinal disorders) | 9 | 1
Injection site reaction (General disorders) | 18 | 6
Influenza (Infections and infestations) | 24 | 6
Nasopharyngitis (Infections and infestations) | 18 | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 5
Headache (Nervous system disorders) | 14 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.